CLINICAL TRIAL: NCT02730338
Title: INTense ExeRcise for SurviVAL Among Men with Metastatic Prostate Cancer (INTERVAL - GAP4): a Multicentre, Randomised, Controlled, Phase III Study
Brief Title: INTense ExeRcise for SurviVAL Among Men with Metastatic Prostate Cancer (INTERVAL - GAP4)
Acronym: INTERVAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Movember Foundation (Other)
Collaborators: University of California, San Francisco (Other); Edith Cowan University (Other); King's College London (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAP4
Record Dates: First submitted 2016-03-10; First posted 2016-04-06 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Prostate Cancer
Keywords: Castrate resistant; Exercise; Metastatic; Prostate cancer; Hormone sensitive
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity; Neoplasm Metastasis | interventions — Resistance Training; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Supervised exercise group (Active Comparator): Supervised high intensity aerobic and resistance exercise tapering to self management with psychosocial support
  Interventions: Behavioral: High intensity aerobic and resistance training; Behavioral: Psychosocial support
- Arm B: Self directed exercise group (Other): Self directed exercise and psychosocial support group
  Interventions: Behavioral: Psychosocial support

INTERVENTIONS:
Behavioral: High intensity aerobic and resistance training
  Arms: Arm A: Supervised exercise group
Behavioral: Psychosocial support

SUMMARY:
To determine if supervised high intensity aerobic and resistance training increases overall survival compared to self-directed exercise in patients with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

mCRPC status:

* mCRPC patients defined as; adenocarcinoma of the prostate with systemic metastatic disease despite castrate levels of testosterone (<50 ng/dL) due to orchiectomy or LHRH agonist.

  o Patients must have one or more of the following to be considered mCRPC
* Metastatic Disease Progression: >20% increase in the sum of diameters of measurable lesions from the time of maximal regression or appearance of one or more new lesions.
* Bone Scan Progression: Appearance of one or more new lesions on bone scan attributable to prostate cancer.
* PSA Progression: PSA ≥2 ng/ml that has risen serially on at least two occasions, each at least one week apart (PSA1 < PSA2 < PSA3).
* PSMA PET/CT scan progression: Appearance of one or more new lesions on PSMA PET/CT scan attributable to prostate cancer.
* At enrolment, mCRPC patients must fit into one of the following 5 categories:

  1. Treatment naïve for mCRPC (have not yet started approved therapies for CRPC ie: Abiraterone/Enzalutamide/Apalutamide / or Docetaxel, Cabazitaxel or other approved first line chemotherapy; less than 4 weeks on approved therapies is still considered to be treatment naïve) Or
  2. Receiving Abi/Enza/Apa for mCRPC AND responding or stable (PSA values must be stable or declining after at least 4 weeks since starting Abi/Enza/Apa for mCRPC) Or
  3. Patients with PSA progression while on Abi/Enza/Apa are eligible as long as they are asymptomatic AND there is no intent on starting chemotherapy within 6 months Or
  4. Patients treated with Docetaxel, Cabazitaxel or other approved first line chemotherapy as first line for mCRPC who are asymptomatic without ANY evidence of progression Or
  5. Patients may have progressed following first line Docetaxel, Cabazitaxel or other first line chemotherapy and are now receiving treatment with Abi/Enza/Apa. These patients must absolutely be responding or stable (PSA values must be stable or declining after starting Abi/Enza/Apa treatment) and have an estimated life expectancy of more than 1 year.

     mHSPC Status:
* mHSPC patients must be classified as either high-risk or high-volume mHSPC. These groups are defined as adenocarcinoma of the prostate with systemic metastatic disease and patients also fit into one of the following 2 categories: 6. High-risk: defined as having at least 2 of three criteria: (i) Gleason score ≥8, (ii) presence of ≥3 lesions on bone scan, or (iii) presence of INTERVAL Protocol Version 5.0, 19 August 2019 4 measurable visceral lesions (PSMA PET imaging should not be used in the definition of high-risk disease) Or 7. High-volume: defined as having the presence of visceral metastases and/or ≥ four bone metastases with at least one outside of the vertebral column and pelvis (PSMA PET imaging should not be used in the definition of high-volume disease)

Additional criteria for all groups:

* All patients will be required to be on ADT during the study period or have had a prior bilateral orchiectomy.
* Men with small cell neuroendocrine tumours or features of small cell disease are not eligible.
* ≥4 weeks since last major surgery and fully recovered.
* No known contraindications to high intensity exercise, including, but not limited to: brain metastases; current congestive heart failure (New York Heart Association Class II, III or IV); serious or non-healing wound, ulcer, or bone fracture; spinal cord compromise or instrumentation due to metastatic disease; peripheral neuropathy ≥grade 3. No serious cardiovascular events within 12 months including, but not limited to, transient ischemic attack (TIA), cerebrovascular accident (CVA), or myocardial infarction (MI). Patients with a history of hypertension must be well-controlled (< 160/90) on anti-hypertensive therapy.
* Halabi Nomogram score <1951 (Risk Category rated as low or intermediate risk)
* Age ≥18 years
* Required Baseline Laboratory Values: ANC ≥ 1500/uL; Platelet count ≥ 100,000/uL; Creatinine ≤ 1.5 x upper limits of normal; Bilirubin ≤ 1.5 x upper limits of normal; AST ≤ 1.5 x upper limits of normal; Serum testosterone ≤ 50 ng/dL
* ECOG performance status 0-1
* Medical clearance by treating physician to undergo a symptom-limited cardiopulmonary exercise test and vigorous aerobic and resistance exercise training, and able to complete an acceptable cardiopulmonary exercise test.
* Exercise Coordination Centre (ECC) review and approval of subject's screening bone scan / areas with bone metastases.
* Men participating in vigorous aerobic exercise for >60 min/week or structured resistance exercise ≥2 days/week, are not eligible.
* Subject is willing and able to use technological aspects of the trial.
* The subject is fluent in the language as designated by the institution at which he would be enrolled.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 866 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | up to 5 years
  Overall survival will be measured from the time of randomization until death

SECONDARY OUTCOMES:
Disease Progression | up to 5 years
  Time to disease progression will be measured from randomization until the first of the following: first CT or bone scan documenting disease progression, initiation of a new therapy for mPC (clinical progression), or first occurrence of a Symptomatic Skeletal Related Event (SSE).
Symptomatic Skeletal Related Events (SSE) | up to 5 years
  Time to first occurrence of SSE will be defined as the time from randomization to documentation of any of the following (whichever occurs first) + 1 day:
  * Use of external beam radiation therapy to relieve bone pain
  * Occurrence of new symptomatic pathological bone fractures that may be vertebral or non-vertebral. Asymptomatic compression fractures detected by radiology review only will not be considered a SSE.
  * Spinal cord compression
  * Change in antineoplastic therapy to treat bone pain
  * Surgical intervention to treat bone pain
Opiate Use | up to 5 years
  Opiate use will be assessed via BPI-SF, the medical record review at entry with a lead-in period (<28 days). The questionnaires will be administered every three cycles until month 24, and in month 36.
Analgesic Use | up to 5 years
  Analgesic use will be assessed via BPI-SF, the World Health Organisation (WHO) analgesic scale, and medical record review at entry with a lead-in period (<28 days). The WHO analgesic scale will be completed every three cycles (based on medical review) and questionnaires will be administered every three cycles until month 24, and in month 36.
Biomarker analysis | up to 5 years
  Inflammatory and cytokine systemic milieu
Biomarker analysis | up to 5 years
  Insulin/Glucose Metabolism
Biomarker analysis | up to 5 years
  Androgen biosynthesis
Quality of Life | up to 5 years
  Physical and emotional quality of life measured by the questionnaires- Functional Assessment of Cancer Therapy- Prostate (FACT-P), Functional assessment of Chronic Illness Therapy (FACIT-Fatigue), and EuroQOL Five Dimension Questionnaire (EQ5D) will be assessed every 3 cycles.
Physical Function | up to 5 years
  Physical function will be assessed using strength assessments (1RM), a cardiopulmonary exercise test (CPET) and a functional performance test (400m walk)
Pain | up to 5 years
  Pain will be assessed via questionnaire Brief Pain Inventory- short form (BPI-SF) and medical record review at entry with a lead-in period (<28 days) and repeated measures will occur every three cycles

CONTACTS AND LOCATIONS:
Overall Officials: Robert Newton, Study Chair — Edith Cowan University; Fred Saad, Study Chair — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (18):
- United States (6):
  - Cedars Sinai Medical Centre, Los Angeles, California
  - UCSF, San Francisco, California
  - UC Denver, Denver, Colorado
  - University of Minnesota, Minneapolis, Minnesota
  - Oregon Health & Science University, Portland, Oregon
  - Fred Hutchinson Cancer Centre, Seattle, Washington
- Australia (4):
  - Australian Prostate Cncr Research Centre, Brisbane, Queensland
  - University of Queensland, Brisbane, Queensland
  - Victoria University / Sunshine Hospital, Melbourne, Victoria
  - Edith Cowan University, Perth, Western Australia
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal
- German Sport University Cologne, Cologne, Germany
- Erasmus MC, Rotterdam, Netherlands
- United Kingdom (4):
  - University of Surrey, Guildford, Surrey
  - Queen's University Belfast, Belfast
  - University of Glasgow, Glasgow
  - Kings College London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Umlauff L, Kenfield SA, Newton RU, Hart NH, Saad F, Courneya KS, Greenwood R, Bloch W; INTERVAL-GAP4 Steering Committee/Coordinating Centres Members/Protocol Development Working Group Members; Schumann M. Meeting Aerobic Physical Activity Guidelines and Associations With Physical Fitness in Men With Metastatic Prostate Cancer: Baseline Results of the Multicentre INTERVAL-GAP4 Trial. Cancer Med. 2024 Dec;13(23):e70261. doi: 10.1002/cam4.70261. PMID 39632499
- [Derived] Kim JS, Taaffe DR, Galvao DA, Clay TD, Redfern AD, Gray ES, Newton RU. Enhancing circulatory myokines and extracellular vesicle uptake with targeted exercise in patients with prostate cancer (the MYEX trial): a single-group crossover study. BMC Cancer. 2024 Jul 1;24(1):784. doi: 10.1186/s12885-024-12530-0. PMID 38951803
- [Derived] Newton RU, Kenfield SA, Hart NH, Chan JM, Courneya KS, Catto J, Finn SP, Greenwood R, Hughes DC, Mucci L, Plymate SR, Praet SFE, Guinan EM, Van Blarigan EL, Casey O, Buzza M, Gledhill S, Zhang L, Galvao DA, Ryan CJ, Saad F. Intense Exercise for Survival among Men with Metastatic Castrate-Resistant Prostate Cancer (INTERVAL-GAP4): a multicentre, randomised, controlled phase III study protocol. BMJ Open. 2018 May 14;8(5):e022899. doi: 10.1136/bmjopen-2018-022899. PMID 29764892